CLINICAL TRIAL: NCT05565027
Title: Efficacy and Safety of Pulmonary Function Analysis With Dynamic Digital Radiography Total Respiratory Cycle Photography in Healthy Volunteers
Brief Title: Efficacy and Safety of Pulmonary Function Analysis With Dynamic Digital Radiography Total Respiratory Cycle Photography
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 202101-02
Record Dates: First submitted 2022-09-30; First posted 2022-10-04 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Healthy Volunteers
Keywords: dynamic digital X-ray; pulmonary function analysis; healthy volunteers

STUDY DESIGN:
Intervention Model Description: The subject stood on the turntable of the instrument and grasped the postural fixator with both hands up. The subjects pinched their nose and breathed through the disposable filter mouthpiece connected to the pneumotachograph, taking care not to leak air at the corners of the mouth. The subjects were instructed to perform tidal breathing, deep inhalation, deep exhalation, etc., and to perform dynamic DR photography and pneumotachograph monitoring simultaneously. At the end of the examination, assist the subjects to leave the examination equipment and re-measure their vital signs.
Masking Description: Lung volume measurements using the test and reference devices were clearly different and could not be blinded to subjects and investigators, so an open trial design was used.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pneumotachograph (Active Comparator): The subject stood on the turntable of the instrument and grasped the postural fixator with both hands up. The subjects pinched their nose and breathed through the disposable filter mouthpiece connected to the pneumotachograph, taking care not to leak air at the corners of the mouth. The subjects were instructed to perform tidal breathing, deep inhalation, deep exhalation, etc., and to monitor lung volume by pneumotachograph.
  Interventions: Device: Pneumotachograph
- Dynamic digital radiography (Experimental): The subject stood on the turntable of the instrument and grasped the postural fixator with both hands up. The subjects pinched their nose and breathed through the disposable filter mouthpiece connected to the pneumotachograph, taking care not to leak air at the corners of the mouth. The subjects were instructed to perform tidal breathing, deep inhalation, deep exhalation, etc., and to monitor lung volume by dynamic digital radiography analysis.
  Interventions: Device: Dynamic digital radiography

INTERVENTIONS:
Device: Dynamic digital radiography — The use of advanced dynamic X-ray photography and acquisition technology can obtain high-definition dynamic lung images of patients throughout the respiratory cycle for analysis.
  Arms: Dynamic digital radiography
Device: Pneumotachograph — The pneumotachograph monitors the flow rate, and the lung volume is calculated by integrating.
  Arms: Pneumotachograph

SUMMARY:
The digital X-ray system produced by Shenzhen Angell Technology Co., Ltd was selected as the tested equipment, and the powerlab biological signal acquisition and analysis system equipped with a pneumotachograph by ADInstruments was selected as the reference equipment. During the study, the lung volume measurements obtained by the lung function analysis method based on the dynamic digital radiography full respiratory cycle photography of the tested equipment was compared with the lung volume measurements obtained by the reference device pneumotachograph. The consistency of the lung volume measurements was used as the main validity evaluation index to observe the distribution of the differences between the measured values of the test device and the reference device, and to verify the validity of the declared product according to the main validity evaluation index.

DETAILED DESCRIPTION:
Pulmonary function test is a test to explore the functional status of human respiratory system with the knowledge of exercise respiratory physiology and modern examination technology. It is an important test content for clinical diagnosis, severity assessment, treatment and prognosis assessment of chest and lung diseases, which has been widely used in the fields of respiratory medicine, surgery and anesthesiology. Compared with chest X-rays and CT examinations, which reflect the static function of the chest and lungs, pulmonary function tests can better reflect the dynamic functional changes of the body.

However, pulmonary function test is not well performed to assess the functional status in patients with poor cooperation (e.g., poor lung function, inability to understand cooperation). Dynamic digital X-ray whole respiratory cycle photography uses advanced dynamic radiography and acquisition technology to obtain high-definition dynamic lung images during the whole respiratory cycle of the patient, and uses the industry's first rotating foot pedal to rotate the patient to obtain weighted 3D scan data and single-angle or multi-angle lung data. The patient's lung function is analyzed by algorithmically extracting the patient's full respiratory cycle airway nodes and branches and data statistics. For patients who cannot cooperate with the lung function, it can provid information on the dynamic function of the patient's chest and lungs for doctors to further improve clinical diagnosis and treatment.

At present, the digital X-ray system (DTP580B-3) and the patient position fixation frame MRW-P1 manufactured by Shenzhen Angell Technology Co., Ltd. have passed the inspection by the inspection agency certified by the State Drug Administration of China (NMPA). Clinical trials were conducted to further evaluate the clinical effectiveness and safety of the products.

The lung volume was measured using a pneumotachograph (with a physiological signal recorder) and a digital X-ray system (UC dynamic DR) in the same healthy subject, and the lung volume values measured by each of the reference device were analyzed for consistency to evaluate the validity of the lung volume measurement by the test device. And To evaluate the safety of the lung volume measurement function of the test device in clinical use based on the occurrence of device malfunctions, adverse events and serious adverse events in the trial.

ELIGIBILITY:
Inclusion Criteria:

① age ≥ 18 years; ② subjects willing to undergo chest radiography; ③ normal pulmonary ventilation function (forced vital capacity (FVC) ≥ 80% of the expected value; forced expiratory volume in first second (FEV1) ≥ 80% of the expected value; 1 second rate (FEV1/FVC) ≥ 70%); ④ can perform tidal breathing, deep inspiration and deep expiration; ⑤ no history of smoking; ⑥ no history of chronic respiratory disease; ⑦ no acute respiratory disease within 4 weeks; ⑧ subjects willing to provide written informed consent

Exclusion Criteria:

① Pregnant and lactating women; ② Inability to stand alone; ③ Severe vertigo and other adverse reactions to rotation in place.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-10-20 (Estimated); Primary Completion 2023-07-20 (Estimated); Study Completion 2023-10-20 (Estimated)

PRIMARY OUTCOMES:
Lung volume changes | 1 day (The start time is when the subject is positioned and begins to breathe on command, and the end time is when the subject safely exits the x-ray system.)
  The volume of gas inhaled/exhaled during each respiratory session of the subject during the monitoring period.

CONTACTS AND LOCATIONS:
Overall Officials: Rongchang Chen, PhD, Study Chair — Shenzhen People's Hospital